CLINICAL TRIAL: NCT05844410
Title: Predictors of All-cause Mortality in Hospitalized COVID-19 Patients Taking Corticosteroids: a Multicenter Retrospective Cross-sectional Study
Brief Title: Evaluation of Corticosteroids Use and Clinical Outcomes in Hospitalized COVID-19 Patients: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Lebanese University (Other)
Responsible Party: Principal Investigator, Georges Hatem, Principal investigator, Lebanese University
Other Study IDs: CRU329
Record Dates: First submitted 2023-05-03; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Pandemic; Morality
MeSH Terms: conditions — COVID-19 | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Corticosteroid — Adults patients admitted to the hospital after a confirmed COVID-19 infection, irrespective of the stage and severity of the disease, were included in the study. Only those receiving corticosteroids as a treatment were in the study sample, with no preferences based on race or ethnicity

SUMMARY:
Despite the recommendations to avoid using corticosteroids systematically for hospitalized coronavirus disease of 2019 (COVID-19) patients, healthcare professionals used personalized treatments, including corticosteroids, as adjuncts to treat their patients due to their limited access to treatment options. This study aims to evaluate the use of corticosteroids among hospitalized COVID-19 patients with all-cause mortality as the primary outcome and to assess the predictors of all-cause mortality associated with the characteristics of the patients and the corticosteroid regimens adopted.

DETAILED DESCRIPTION:
A multicenter retrospective study was performed over three months targeting 422 COVID-19 patients from six hospitals in Lebanon. Data were collected from patients' medical charts retrospectively and covered a period of one year (September 2020 to August 2021). The study sample included 422 patients, predominantly males, with 59% of cases classified as severe or critical cases. Dexamethasone and methylprednisolone were the most used corticosteroids. Around 22% of the patients died during hospitalization. After adjusting for covariates, performing a polymerase chain reaction test before admission increased the mortality rate by 424% compared to doing it at hospital admission (adjusted Hazard Ratio (aHR) 4.24, 95% Confidence Interval (CI) 1.35-13.3), with 18.11 times higher mortality rate among critical cases (aHR 18.11, 95% CI 9.63-31.05). Exposure to side effects from corticosteroids increased the mortality rate by 514% compared to others (aHR 5.14, 95% CI 1.28-8.58). In particular, the mortality rate among patients having hyperglycemia dropped by 73% compared to others (aHR 0.27, 95% CI 0.06-0.98). Corticosteroids are frequently used in treating hospitalized COVID-19 patients. The all-cause mortality rate was higher among older and critical cases and lower among smokers and those treated for more than 7 days. Research exploring the safety and efficacy of corticosteroids is required to allow better in-hospital management of COVID-19 cases.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients admitted to the hospital after a confirmed COVID-19 infection, irrespective of the stage and severity of the disease, were included in the study.

Exclusion Criteria:

* Only those receiving corticosteroids as a treatment were in the study sample, with no preferences based on race or ethnicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients admitted to the hospital after a confirmed COVID-19 infection, irrespective of the stage and severity of the disease, were included in the study.
Sampling Method: Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Lebanese University Faculty of pharmacy, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided